CLINICAL TRIAL: NCT03572738
Title: Hidradenitis Suppurativa Mail Survey
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00049730
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa
Keywords: acne inversa; HS; Verneuil's Disease
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HS: The set of all Hidradenitis Suppurativa patients (ICD-10 code: L73.2) who visited Wake Forest Baptist Medical Center's dermatology clinic during the last 5 years will either be recruited in person or be mailed the HS Severity Self-Assessment tool and a survey about their demographics, symptoms, treatments, psychological aspects, and lifestyle.

SUMMARY:
Hidradenitis Suppurativa (HS), also known as "acne inversa," is a chronic dermatologic disease affecting apocrine gland-bearing areas and presenting with symptoms ranging from pustules and inflammatory nodules to draining sinuses, abscesses, and fistulae. The pain and odorous lesions associated with HS contribute to its heightened impact on quality of life in comparison to other diseases; it has been described as "one of the most distressing conditions observed in dermatology." Though it is clear that HS has a significant impact on quality of life, how this manifests remains poorly characterized. The aim of this study is to characterize the quality of life impact of HS and to validate a tool for patients to self-assess the severity of their condition.

DETAILED DESCRIPTION:
Running a comprehensive study and asking patients what challenges they encounter in their daily lives can shed light on the ways in which HS causes quality of life impairment. In this study, the study team aims to identify the following: problems faced by patients with HS, the rate of depression, the rate of stigmatization, the rate of fear of being accepted in society, treatments that patients have tried (and which treatments seem to have worked best), the rate of alternative treatment use, and the correlation of these factors with the severity of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Hidradenitis Suppurativa by a dermatologist at Wake Forest Baptist Medical Center's dermatology clinic.
* Patients 18 years of age or older

Exclusion Criteria:

* Patients younger than 18 years of age
* Any patient who does not have a mailing address on file

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subset of all Hidradenitis Suppurativa patients who visited the Wake Forest Baptist Medical Center's dermatology clinic during last 5 years will be mailed questionnaires and recruited in clinic.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Comparison of self-assessed severity to physician-assessed severity of HS | 1 day
  Participants will be administered a 2-page survey with photographs of HS in varying degrees of severity (Hidradenitis Suppurativa Self-Assessment tool, or HSSA) and asked to check the photo(s) that represent their condition now and when it was the worst it has ever been. The photos correspond with severity levels 0 (no disease), 1, 2, and 3 according to the Hurley Staging system (a commonly used system to evaluate severity of HS). Physicians will also assess the Hurley severity of disease when they see the patient. Agreement between physician severity assessment and self assessment will be measured.
Test-retest reliability of self-assessed severity of HS | 1 day
  Participants will be administered a 2-page survey with photographs of HS in varying degrees of severity and asked to check the photo(s) that represent their condition now and when it was the worst it has ever been. The photos correspond with severity levels 0 (no disease), 1, 2, and 3 according to the Hurley Staging system (a commonly used system to evaluate severity of HS). At least 30 minutes later, participant's will re-do the HSSA. Agreement between the original and second response will be assessed to establish test-retest reliability of the tool.
Ability of HSSA to detect changes in disease severity over time | 1 day
  For those patients who are recruited in person, when they come back to the clinic for follow-up, the HSSA will be administered again. The physician will also provide an assessment of severity. These will be compared to the original physician assessment and HSSA result to determine the ability of the HSSA to detect changes in disease severity over time.

SECONDARY OUTCOMES:
Quality of life as measured by DLQI | 1 day
  Patients will be administered a survey either in clinic or by mail that includes several baseline characteristics and metrics. The Dermatology Life Quality Index (Finlay and Khan) is one of these metrics; it is a standardized questionnaire assessing a patient's quality of life. This will be scored according to standard guidelines and assessed in all subjects. The scores range from 0 to 30, with a higher score indicating higher quality of life impairment. Further analysis may be done to group quality of life by severity and baseline characteristics.
Quality of life as measured by HiSQoL | 1 day
  Patients will be administered a survey either in clinic or by mail that includes several baseline characteristics and metrics. The Hidradenitis Suppurativa Quality of Life survey (McLellan, Sisic, Oon, Tan) is one of these metrics; it is a standardized questionnaire assessing a patient's quality of life. This will be scored according to standard guidelines and assessed in all subjects. Each factor is rated on a scale from 0-4, 0 meaning HS does not influence that factor at all, and 4 meaning the factor is affected greatly by HS. Thus, higher numbers correlate with higher quality of life impact. Further analysis may be done to group quality of life by severity and baseline characteristics.
Quality of life as measured by RAND-36 | 1 day
  Patients will be administered a survey either in clinic or by mail that includes several baseline characteristics and metrics. The RAND-36 is one of these metrics; it is a standardized questionnaire assessing a patient's quality of life. This will be scored according to standard guidelines and assessed in all subjects. In terms of scoring, questions are grouped into broader categories: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health, and health change. Each group is assigned a percentage based on responses (0-100), and a higher percentage signifies better quality of life for each category (the greatest is 100%). Further analysis may be done to group quality of life by severity and baseline characteristics.
Depression as measured by PHQ-9 | 1 day
  Patients will be administered a survey either in clinic or by mail that includes several baseline characteristics and metrics. The PHQ-9 is one of these metrics; it is a standardized questionnaire assessing severity of depression. This will be scored according to standard guidelines and assessed in all subjects. For each of the 9 questions, scores can range from 0-3, 3 being the worst (experiencing the symptom nearly every day). These numbers are summed. A score of 0-4 signifies no depression, 5-9 signifies mild depression, 10-14 signifies moderate depression, 15-19 signifies moderately severe depression, and 20-27 signifies severe depression. Further analysis may be done to group depression status by severity of HS and baseline characteristics.
Fear of Negative Evaluation | 1 day
  Patients will be administered a survey either in clinic or by mail that includes several baseline characteristics and metrics. The Brief Fear of Negative Evaluation survey (Leary) is one of these metrics; it is a standardized questionnaire assessing social anxiety. This will be scored according to standard guidelines and assessed in all subjects. The score for each question ranges from 0-5, and 4/12 items are reverse coded. Higher scores indicated higher levels of social anxiety. Further analysis may be done to group scores by severity and baseline characteristics.
Emotional Stability as measured by PANAS (Positive and Negative Affect Schedule) | 1 day
  Patients will be administered a survey either in clinic or by mail that includes several baseline characteristics and metrics. The PANAS is one of these metrics; it is a standardized questionnaire assessing levels of positive and negative affect. This will be scored according to standard guidelines and assessed in all subjects. The PANAS consists of 20 questions. 10 questions measure positive affect, with scores ranging from 10-50 and higher scores indicating greater positive affect. Similarly, 10 questions measure negative affect, with scores ranging from 10-50, with smaller scores indicating lower levels of negative affect. Further analysis may be done to group scores by severity and baseline characteristics.
Stigmatization as measured by an adaptation of Ginsburg and Link Feelings of Stigmatization | 1 day
  Patients will be administered a survey either in clinic or by mail that includes several baseline characteristics and metrics. The Feelings of Stigmatization survey (adapted from Ginsburg and Link) is one of these metrics; it is a standardized questionnaire assessing stigma associated with disease. This will be scored according to standard guidelines and assessed in all subjects. The adapted survey contains 31 questions asking about stigmatization. Aside from the reverse coded questions, higher scores indicate greater levels of stigmatization (for each question, the score ranges from strongly agree to strongly disagree). Further analysis may be done to group scores by severity and baseline characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Feldman, M.D., Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ball SL, Tidman MJ. Managing patients with hidradenitis suppurativa. Practitioner. 2016 May;260(1793):25-9, 3. PMID 27382916
- [Background] Wolkenstein P, Loundou A, Barrau K, Auquier P, Revuz J; Quality of Life Group of the French Society of Dermatology. Quality of life impairment in hidradenitis suppurativa: a study of 61 cases. J Am Acad Dermatol. 2007 Apr;56(4):621-3. doi: 10.1016/j.jaad.2006.08.061. Epub 2006 Oct 20. PMID 17097366
- [Background] Alavi A, Anooshirvani N, Kim WB, Coutts P, Sibbald RG. Quality-of-life impairment in patients with hidradenitis suppurativa: a Canadian study. Am J Clin Dermatol. 2015 Feb;16(1):61-5. doi: 10.1007/s40257-014-0105-5. PMID 25432664